CLINICAL TRIAL: NCT02974114
Title: Assessment of Cognitive Function and Mobility in Individuals With Pain
Brief Title: Exploratory Study to Investigate Cognition Function and Mobility in Individuals With Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 204503
Record Dates: First submitted 2016-09-19; First posted 2016-11-28 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Paracetamol and caffeine (Experimental): Participants will be administered test product (containing 500 mg paracetamol and 65 mg caffeine). Two tablets will be taken orally once with 200 mL (milliliters) of water.
  Interventions: Drug: Paracetamol and caffeine
- Paracetamol (Experimental): Participants will be administered test product (containing 500 mg paracetamol). Two tablets will be taken orally once with 200 mL of water.
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Participants will be administered reference product (placebo to match Paracetamol 665mg sustained release tablets). Two tablets will be taken orally once with 200 mL of water.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Paracetamol and caffeine — Test product containing 500 mg paracetamol and 65 mg caffeine
  Arms: Paracetamol and caffeine
Drug: Paracetamol — Test product containing 500 mg paracetamol
  Arms: Paracetamol
Other: Placebo — Placebo to match paracetamol 665mg sustained release tablets
  Arms: Placebo

SUMMARY:
This parallel, assessor blind, placebo-controlled, stratified, randomized study will investigate the effects of everyday pain on cognition and mobility in otherwise healthy individuals.

DETAILED DESCRIPTION:
This study consisted of 3 visits. Visit 1 (Day1, Screening), minimum (min) of 7 days and maximum (max) of 28 days gap followed by Visit 2 (Day 2, pain-state assessment), a recovery period of min of 2 days and max of 30 days followed by Visit 3 (Day 3, pain-free assessment). Participants received treatment once only on Visit 2.

ELIGIBILITY:
Inclusion Criteria

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Aged between 18-65 years.
* Participant is male or female.
* Understands and is willing, able and likely to comply with all study procedures and restrictions.
* Adequately completes cognition and mobility familiarisation tasks in the opinion of the investigator.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon physical examination; absence of any condition that might impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements; BMI >18.5 and <30 kg/m2
* VISIT 1 ONLY - Has experienced a minimum of two recurrent, acute pain episodes within the past 3 months or is currently suffering from a flare up episode of recurrent, acute pain; VISIT 2 ONLY - A score ≥5 to question 6 (rated on scale 0-10) on the Brief Pain Inventory - Short Form and participants presenting with only one of the following pain types: Joint (Knee, Hip); Back; Headache; Period.

Exclusion Criteria

* Women who are pregnant (Visit 1), women of child bearing potential who test positive on a urine pregnancy test (Visit 1 or Visit 2), females of non-child bearing potential will not be required to complete urinary pregnancy test, post-menopausal females not requiring a pregnancy test will be defined as: Age ≥ 50 years with spontaneous cessation of menses for 12 or more months or age < 55 years and spontaneous menses within the past 1 year, but currently amenorrheic.
* Women who are currently breast-feeding.
* In the opinion of the medical designee, participant suffers from medical condition(s) that may be aggravated due to testing procedures or may impact the interpretation or integrity of data. Conditions related to renal, hepatic, respiratory, blood, immune systems or heart dysfunction will be considered.
* Participant is colour blind.
* Current (within 14 days of the start of the study) or regular use of any prescription, over-the-counter (OTC), herbal medicine unless the medication has been approved by the study physician. OTC analgesics for pain relief and vitamin supplements are permitted only until 48 hours prior to study visits; Current or in the 30 days prior to dosing use of any drug, food, herbal product, or dietary supplement known to induce or inhibit hepatic drug metabolism (e.g. barbiturates, theophylline, cimetidine, or erythromycin) ;Use of analgesics and anti-inflammatory drugs 48 hours prior to dosing at Visit 2; Known to be taking any other medication which could counteract with paracetamol and/or caffeine; Current or past use of anti-depressants or psychoactive drugs within the previous 2-years.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Positive breath alcohol test at Visit 2 and positive urine drugs of abuse test at Visit 2.
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational product within 7 days of the screening visit or previous participation and randomization in this study.
* Participant has excessive frequent caffeine intake equivalent to 6 cups of brewed coffee or 12 cups of tea per day; Unwilling to abstain from any caffeine products from 4 hours prior to the visit on assessment days (Visit 2 and 3); Current Smoker (or regular nicotine consumption): Participant smokes more than 3 cigarettes per day (or equivalent for e-cigarettes, chewing tobacco or pipes). Investigator will ensure there is no impact of withdrawal effect from those with nicotine dependence; Current Alcohol Consumer: Participant consumes greater than 21 units of alcohol per week (male) and 14 units per week (female) (e.g. Spirit 25ml = 1 unit / AlcoPop 275ml = 1.5 unit / Bottle of beer 330 ml = 1.7 unit / Glass of wine 175ml = 2.1 unit / Pint of beer 568 ml = 3 unit).
* Members of the study site staff or members of their immediate family.
* Any participant who in the opinion of the investigator should not take part in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Brentford, Middlesex, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited at a single center from the United Kingdom.
Pre-assignment Details: A Total of 54 participants were screened, out of which 21 participants were randomized to the study, 5 participants were screening failure, 1 participant withdrew consent and 27 participants were not randomized due to other reasons (not specified).
Groups:
- Paracetamol and Caffeine: All the participants in this arm received test product (containing 500 milligram [mg] of paracetamol and 65 mg of caffeine). All the participants took 2 tablets at once orally with 200 milliliters (mL) of water.
- Paracetamol: All the participants in this arm received test product (containing 500 mg of paracetamol). All the participants took 2 tablets orally once with 200 mL of water.
- Placebo: All the participants in this arm received reference product (placebo to match Paracetamol 665mg sustained release tablets). All the participants took 2 tablets orally once with 200 mL of water.
Period: Overall Study
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Started | 6 | 7 | 8
Completed | 6 | 6 | 6
Not Completed | 0 | 1 | 2
Not completed — Other (Not specified) | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Paracetamol and Caffeine: All the participants in this arm received test product (containing 500 mg of paracetamol and 65 mg of caffeine). All the participants took 2 tablets orally once with 200 mL of water.
- Total: Total of all reporting groups
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.8 (4.83) | 30.0 (9.45) | 40.0 (15.87) | 33.2 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 2 | 2 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 3 | 5 | 4 | 12
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Pain Free State (Day 3) in Error Adjusted Simple Reaction Time (SRT) in the Pain State (Day 2)
Description: Error adjusted SRT was one of the main outcomes of the Axon Sports Priming Application. The Axon Sports Priming Application is a computerized test performed on a tablet device that measures cognitive performance, namely psychomotor speed. Axon sports test assessment included 1. Pain-state assessment performed at Visit 2 (Day 2 pre-treatment assessment and post-treatment assessment 1hour [hr] ± 15 minutes [mins] post-dosing) and 2. Pain-free assessment performed at Visit 3 (Day 3).
Time Frame: At Day 2 (pre and post-treatment) and Day 3 of the study
Population: Modified Intent-to-Treat (mITT, N=20) Population: All the participants who were randomized, received at least one dose of the study treatment and had at least one post-baseline assessment without any violation of study inclusion-exclusion criteria were included in the mITT population.
Measure: Median (Full Range); unit: milliseconds (msec)
Groups:
- Paracetamol and Caffeine: All the participants in this arm received test product (containing 500 mg of paracetamol and 65 mg of caffeine). All the participants took 2 tablets at once orally with 200 mL of water.
- Paracetamol: All the participants in this arm received test product (containing 500 mg of paracetamol). All the participants took 2 tablets at once orally with 200 mL of water.
- Placebo: All the participants in this arm received reference product (placebo to match Paracetamol 665mg sustained release tablets). All the participants took 2 tablets at once orally with 200 mL of water.
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
milliseconds (msec)
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | 0.05 [0.0 to 0.2] | 0.07 [0.0 to 0.8] | 0.06 [0.0 to 0.2]
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | 0.04 [0.0 to 0.4] | 0.01 [0.0 to 0.3] | 0.00 [-0.2 to 0.1]

2. Primary Outcome: Change From Pain-free State (Day 3) in Reaction Time in the Pain State (Day 2)
Description: The reaction time of five-choice reaction time task (provided by Cambridge Cognition) was measured. In five-choice reaction time task, all the participants hold down a button at the bottom of the screen till a yellow spot appears in one of the five circles at the top of the screen. Participants then released the button and touch inside of the circle where the yellow spot appeared as quickly as they can. The median duration, between the onset of the stimulus and the release of the button, was recorded as reaction time. Calculated for correct, assessed trials where the stimulus appeared in any one of five locations.
Time Frame: At Day 2 (pre and post-treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Median (Full Range); unit: msec
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
msec
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | 2.00 [-17.5 to 36.0] | -1.75 [-41.0 to 170.5] | -1.00 [-6.5 to 18.5]
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | 25.75 [-11.5 to 83.5] | 12.50 [-65.5 to 26.0] | -8.00 [-28.0 to 24.5]

3. Primary Outcome: Change From Pain-free State (Day 3) in Number of One Touch Stockings (OTS) of Cambridge Assessment Problems (on Which the First Box Choice Made Was Correct) in the Pain State (Day 2)
Description: OTS was a measure of executive function and takes approximately 10 minutes to complete. The participant was shown two displays containing three coloured balls. The displays were presented in such a way that they can easily be perceived as stacks of coloured balls held in stockings or socks suspended from a beam. There was a row of numbered boxes along the bottom of the screen. The test administrator first demonstrated to the participant how to use the balls in the lower display to copy the pattern in the upper display, and completed one demonstration problem, where the solution requires one move. The participant then completed three further problems, one each of two moves, three moves, and four moves. Next, the participant was shown further problems, and participants worked out in their head how many moves the solutions to these problems required, and then touch the appropriate box at the bottom of the screen to indicate their response.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: OTS of correct first box choice
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
OTS of correct first box choice
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | -2.67 (3.077) | 0.00 (1.095) | -0.20 (1.789)
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | -1.83 (1.941) | 2.17 (1.835) | -1.40 (2.702)

4. Primary Outcome: Change From Pain-free State (Day 3) in Attention Switching Task (AST) Congruency Cost in the Pain State (Day 2)
Description: AST was a measure of executive attention. The test displayed an arrow which can appear on either side of the screen and can point in either direction. Each trial displayed a cue at the top of the screen that indicates whether to press the right or left button. Some trials displayed congruent stimuli (e.g. arrow on the right side of the screen pointing to the right) whereas other trials display incongruent stimuli which require a higher cognitive demand (e.g. arrow on the right side of the screen pointing to the left). The AST congruency cost was the difference between the median latencies of response (from stimulus appearance to button press) on the trials that were congruent versus the trials that were incongruent. It was calculated by subtracting the median of congruent from incongruent latency. A positive score indicated response was faster on congruent trials and a negative score indicated response was faster on incongruent trials.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Median (Full Range); unit: msec
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
msec
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | -3.25 [-44.5 to 46.5] | 46.25 [-22.5 to 99.5] | 2.50 [-4.0 to 113.5]
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | -8.25 [-44.0 to 43.5] | 23.00 [-5.0 to 104.0] | 22.50 [-171.5 to 113.5]

5. Primary Outcome: Change From Pain-free State (Day 3) in Spatial Working Memory (SWM) Between Errors in the Pain State (Day 2)
Description: SWM task was a measure of working memory. The task involved number of coloured squares (boxes) being shown on the screen. The aim of this test was to find one blue token in the boxes shown to the participants by process of elimination and used these to fill up an empty column on the right-hand side of the screen. The number of boxes gradually increased up to a maximum of eight boxes to search and the colour and position of the boxes changed from trial to trial. SWM between errors was defined as times the participant revisited a box in which a token has previously been found. This was calculated for trials of four, six and eight tokens.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SWM between errors
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
SWM between errors
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | -9.33 (18.747) | 25.17 (29.075) | 13.80 (23.994)
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | 4.83 (22.248) | 13.50 (23.193) | -9.80 (32.920)

6. Primary Outcome: Change From Pain-free State (Day 3) in Rapid Visual Information Processing A Prime (RVPA) in the Pain State (Day 2)
Description: RVP task was measures of attention. A white box appeared in the centre of the computer screen, inside which digits, from 2 to 9, appeared in a pseudo-random order, at the rate of 100 digits per minute. Participants were requested to detect target sequences of digits (for example, 2-4-6, 3-5-7, 4-6-8) and to register responses using the press pad. The RVPA (A prime) was the signal detection measure of sensitivity to the target, regardless of response tendency (the expected range will be 0.00 to 1.00; bad to good). RVP metric was a measure of how good the subject was at detecting target sequences.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Median (Full Range); unit: msec
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
msec
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 4
  Change from pain-free state at Day 2 pre-treatment | -0.04 [-0.1 to 0.0] | 0.00 [0.0 to 0.0] | -0.03 [-0.1 to 0.0]
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 4
  Change from pain-free state at Day2 post-treatment | -0.02 [-0.1 to 0.0] | -0.01 [-0.1 to 0.0] | 0.00 [0.0 to 0.0]

7. Secondary Outcome: Change From Pain-free State (Day 3) in Grip Force in Pain State (Day 2)
Description: This task was a measure of grip strength. The participant held the dynamometer in their dominant hand and the arm was swung from above the head to by the side of the body. If the dominant arm or hand was painful then the non-dominant hand was used. The participant was instructed to assert maximum effort during the squeezing motion and maintain it for about 4 seconds using a metronome. Participant conducted the movement 4-times (1 practice effort and 3 test efforts) and there was a 1-minute recovery period between each effort.
Time Frame: At Day 2 (pre and post-treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
Kilogram (Kg)
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | -1.98 (5.505) | -3.87 (3.792) | -1.70 (3.533)
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | 0.68 (2.384) | -2.80 (3.059) | -0.46 (1.365)

8. Secondary Outcome: Change From Pain-free State (Day 3) in Time to Standing in Pain State (Day 2)
Description: Time to standing provides a simple assessment of physical mobility. From a seated position with arms crossed so that the right hand is placed on the left shoulder and the left hand on the right shoulder, participants stood to a fully erect stature in as short a time as possible. Time to standing recorded which was measured using a stopwatch. Participants conducted the same movement 3-times continuously as a practice effort and 5-times continuously as a test effort at each visit. There was a 1-minute rest between the practice and test effort.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Median (Full Range); unit: Seconds
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
Seconds
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | 0.10 [-0.4 to 0.2] | 0.13 [-0.2 to 0.3] | 0.09 [0.0 to 0.3]
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | -0.01 [-0.2 to 0.5] | -0.08 [-0.3 to 0.4] | 0.04 [-0.2 to 0.6]

9. Secondary Outcome: Change From Pain-free State (Day 3) in Ground Reaction Force (GRF) in Pain State (Day 2)
Description: From a seated position with arms crossed so that the right hand is placed on the left shoulder and the left hand on the right shoulder, participants stood to a fully erect stature in as short a time as possible. Participants conducted the same movement 3-times continuously as a practice effort and 5-times continuously as a test effort at each visit. There was a 1-minute rest between the practice and test effort. GRF was measured during the movement analyzed using a force plate interfaced with a computer.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
Newtons
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | 3.35 (11.781) | -19.80 (43.788) | 3.75 (11.214)
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | 4.21 (8.295) | -13.85 (47.387) | 3.08 (12.064)

10. Secondary Outcome: Change From Pain-free State (Day 3) in Contact Phase in Pain State (Day 2)
Description: Participants performed a walking assessment in comfortable walking shoes to measure gait parameter contact phase. An athletic movement analysis system (Optojump, Microgate) was utilized which set up over a 15 meters (m) length of track with only the 5-10m section measured and analysed. Participants were instructed to walk the 15m length a minimum of 6 times (3 practice and a minimum of 3 test walks) always entering the 15m length with the same foot first. The foot (left or right) entering the 5-10m section first was recorded by visual assessment of the Optojump operator for the test walks. Test walks were repeated until there were 3 walks in which the participants have entered the 5-10m section with the same foot first.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Median (Full Range); unit: Seconds
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
Seconds
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | 0.03 [0.0 to 0.1] | 0.03 [0.0 to 0.1] | 0.00 [0.0 to 0.0]
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | 0.03 [-0.0 to 0.1] | 0.02 [-0.0 to 0.1] | 0.01 [-0.02 to 0.03]

11. Secondary Outcome: Change From Pain-free State (Day 3) in Stride Length in Pain State (Day 2)
Description: Participants performed a walking assessment in comfortable walking shoes to measure gait parameter stride length. An athletic movement analysis system (Optojump, Microgate) was utilized which set up over a 15 meters (m) length of track with only the 5-10m section measured and analysed. Participants were instructed to walk the 15m length a minimum of 6 times (3 practice and a minimum of 3 test walks) always entering the 15m length with the same foot first. The foot (left or right) entering the 5-10m section first was recorded by visual assessment of the Optojump operator for the test walks. Test walks were repeated until there were 3 walks in which the participants have entered the 5-10m section with the same foot first.
Time Frame: At Day 2 (pre and post treatment) and Day 3 of the study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
Centimeter
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | -0.06 (0.098) | -0.08 (0.123) | -0.02 (0.038)
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | -0.04 (0.084) | -0.06 (0.116) | -0.04 (0.037)

12. Secondary Outcome: Change From Pain-free State (Day 3) in Walking Speed in Pain State (Day 2)
Description: Participants performed a walking assessment in comfortable walking shoes to measure gait parameter walking speed over 5-10m for each foot. An athletic movement analysis system (Optojump, Microgate) was utilized which set up over a 15 meters (m) length of track with only the 5-10m section measured and analysed. Participants were instructed to walk the 15m length a minimum of 6 times (3 practice and a minimum of 3 test walks) always entering the 15m length with the same foot first. The foot (left or right) entering the 5-10m section first was recorded by visual assessment of the Optojump operator for the test walks. Test walks were repeated until there were 3 walks in which the participants have entered the 5-10m section with the same foot first.
Time Frame: At Day 2 (pre and post-treatment) and Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters/second
Groups:
- Paracetamol: All the participants in this arm received test product (containing 500 mg of paracetamol). All the participants took 2 tablets at once orally with 200 milliliters (mL) of water.
- Placebo: All the participants in this arm received reference product (placebo to match Paracetamol 665mg sustained release tablets). All the participants took 2 tablets at once orally with 200 milliliters (mL) of water.
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
Number analyzed (Participants) | 6 | 7 | 7
meters/second
  Change from pain-free state at Day 2 pre-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day 2 pre-treatment | -0.11 (0.112) | -0.10 (0.180) | -0.02 (0.052)
  Change from pain-free state at Day2 post-treatment: number analyzed (Participants) | 6 | 6 | 5
  Change from pain-free state at Day2 post-treatment | -0.10 (0.105) | -0.07 (0.157) | -0.03 (0.043)

ADVERSE EVENTS:
Time Frame: Up to 61 days
Arm/Group | Paracetamol and Caffeine | Paracetamol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 1/7 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paracetamol and Caffeine (N=6) | Paracetamol (N=7) | Placebo (N=8)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to breaches of GCP guidelines observed during a GSKCH internal audit. The minimum requirement of 8 subjects per strata was not met because of early termination so some exploratory analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT02974114/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT02974114/SAP_001.pdf